CLINICAL TRIAL: NCT04502030
Title: Double-blind, Randomized, Placebo-controlled, Prospective Phase III Study Evaluating Efficacy and Safety of Panzyga in Primary Infection Prophylaxis in Patients With Chronic Lymphocytic Leukemia ("PRO-SID" Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NGAM-12
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Chronic Lymphocytic Leukemia; Hypogammaglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Agammaglobulinemia | interventions — Panzyga

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Panzyga (Experimental)
  Interventions: Biological: Panzyga
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Panzyga — Panzyga is a 10% IVIG produced from a pool of human fresh frozen plasma donations
  Arms: Panzyga
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Study Evaluating Efficacy and Safety of Panzyga in Primary Infection Prophylaxis in Patients with Chronic Lymphocytic Leukemia

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-naïve or relapsed/refractory CLL patients undergoing CLL antineoplastic treatment. Diagnosis of B-cell CLL established according to International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria and documented within medical records.
2. Hypogammaglobulinemia (IgG levels <5 g/L) as confirmed by the Central Laboratory.
3. ≥18 years of age.
4. Voluntarily given, fully informed written and signed consent obtained before any study-related procedures are conducted.

Exclusion Criteria:

1. IgG treatment within 3 months prior to Screening.
2. Antibiotic prophylaxis and/or treatment within 7 days prior to Baseline (with the exception of trimethoprim-sulfamethoxazole [TMP/SMX], diaminodiphenyl sulfone [dapsone] and pentamidine inhalation).
3. Current major infection or >1 major infection in the previous 6 months before Baseline.
4. History of anaphylaxis or severe systemic response to immunoglobulin, blood or plasma-derived products or any Panzyga component.
5. History of a non-CLL malignancy or other medical condition with life-expectancy of less than two years.
6. Severe liver disease, with signs of ascites and/or hepatic encephalopathy.
7. Severe kidney disease (as defined by estimated glomerular filtration rate [eGFR] <30 mL/min/1.73 m2).
8. Body weight >140 kg.
9. Eastern Cooperative Oncology Group (ECOG) performance score of >2 (Appendix 1).
10. Female patients of childbearing potential unwilling to use a protocol-required method of contraception (as per protocol section 7.3.9 b) from the Screening Visit throughout the study treatment period and for 30 days following the last dose of study drug.
11. Human immunodeficiency virus (HIV) infection at Screening (defined for the study as positive HIV antibody test).
12. Patients found to be chronic carriers of hepatitis B virus (HBV), defined by positive surface antigen (HBsAg), positive Hepatitis B core antibodies (HBcAb) and/or low HBV titers, who will not receive targeted antiviral therapy while undergoing CLL therapy, and patients with active HBV, defined as high HBV titers.
13. Uncontrolled hepatitis C infection at Screening (defined for the study as positive hepatitis virus C [HCV] polymerase chain reaction [PCR]).
14. Pregnant and lactating women.
15. Subjects with a history of thromboembolic events (TEE) such as deep vein thrombosis, pulmonary embolism, myocardial infarction, ischemic stroke, transient ischemic attack, peripheral artery disease (Fontaine IV) within 6 months before Baseline.
16. Planned or ongoing immunosuppressive treatment (other than for CLL or corticosteroids) or other forbidden medication during the entire study duration after study enrollment.
17. Participation in another interventional clinical trial that is either blinded or involves an investigational (not approved) product within 3 months before Baseline or during the course of the clinical study. Participation in observational clinical trials or open-label trials involving an approved product may be permitted after consultation with the medical monitor.
18. Known IgA deficiency with antibodies to IgA.
19. Known blood hyperviscosity, or other hypercoagulable states.
20. Patients unable or unwilling to understand or comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of major infections | 52 weeks
  Major infection for this trial is defined as:
  * Bacterial and/or viral infections resulting in death
  * Bacterial and/or viral infections, which are microbiologically documented (MDI) or clinically documented (CDI) requiring treatment with anti-infectives; upper respiratory tract infections, bronchitis, lower urinary tract infections, localized skin infections and stomatitis (MDI or CDI) are considered major only if they require treatment with antiinfectives AND hospitalization or hospitalization prolongation.
  * Fever of unknown origin (FUO) requiring hospitalization or hospitalization prolongation

SECONDARY OUTCOMES:
Overall infection rate | 52 weeks
  Infection rate for all infections
Frequency of prophylaxis with anti-infectives | 52 weeks
  Inclusive of antibacterials and antivirals
Duration of prophylaxis with anti-infectives | 52 weeks
  Inclusive of antibacterials and antivirals

CONTACTS AND LOCATIONS:
Locations (74):
- United States (13):
  - Octapharma Research Site, St. Petersburg, Florida
  - Octapharma Research Site, Columbus, Georgia
  - Octapharma Research Site, Macon, Georgia
  - Octapharma Research Site, New Orleans, Louisiana
  - Octapharma Research Site, Baltimore, Maryland
  - Octapharma Research Site, Detroit, Michigan
  - Octapharma Research Site, Rochester, Minnesota
  - Octapharma Research Site, Buffalo, New York
  - Octapharma Research Site, New York, New York
  - Octapharma Research Site, Shirley, New York
  - Octapharma Research Site, Durham, North Carolina
  - Octapharma Research Site, Charleston, South Carolina
  - Octapharma Research Site, Houston, Texas
- Czechia (3):
  - Octapharma Research Site, Brno
  - Octapharma Research Site, Hradec Králové
  - Octapharma Research Site, Ostrava
- Denmark (3):
  - Octapharma Research Site, Aalborg
  - Octapharma Research Site, Herning
  - Octapharma Research Site, Roskilde
- Germany (4):
  - Octapharma Research Site, Dortmund
  - Octapharma Research Site, Frankfurt
  - Octapharma Research Site, Kiel
  - Octapharma Research Site, Marburg
- Greece (4):
  - Octapharma Research Site, Athens
  - Octapharma Research Site, Ioannina
  - Octapharma Research Site, Pátrai
  - Octapharma Research Site, Thessaloniki
- Hungary (5):
  - Octapharma Research Site, Budapest
  - Octapharma Research Site, Debrecen
  - Octapharma Research Site, Győr
  - Octapharma Research Site, Kaposvár
  - Octapharma Research Site, Nyíregyháza
- Israel (2):
  - Octapharma Research Site, Haifa
  - Octapharma Research Site, Petah Tikva
- Italy (9):
  - Octapharma Research Site, Castelfranco Veneto
  - Octapharma Research Site, Milan
  - Octapharma Research Site, Modena
  - Octapharma Research Site, Orbassano
  - Octapharma Research Site, Padua
  - Octapharma Research Site, Pescara
  - Octapharma Research Site, Reggio Calabria
  - Octapharma Research Site, Rome
  - Octapharma Research Site, Torino
- Poland (10):
  - Octapharma Research Site, Bialystok
  - Octapharma Research Site, Bydgoszcz
  - Octapharma Research Site, Gdansk
  - Octapharma Research Site, Gdynia
  - Octapharma Research Site, Katowice
  - Octapharma Research Site, Legnica
  - Octapharma Research Site, Lodz
  - Octapharma Research Site, Torun
  - Octapharma Research Site, Warsaw
  - Octapharma Research Site, Wroclaw
- Russia (13):
  - Octapharma Research Site, Barnaul
  - Octapharma Research Site, Kemerovo
  - Octapharma Research Site, Moscow
  - Octapharma Research Site, Nizhny Novgorod
  - Octapharma Research Site, Novosibirsk
  - Octapharma Research Site, Petrozavodsk
  - Octapharma Research Site, Rostov-on-Don
  - Octapharma Research Site, Saint Petersburg
  - Octapharma Research Site, Samara
  - Octapharma Research Site, Tomsk
  - Octapharma Research Site, Tula
  - Octapharma Research Site, Ufa
  - Octapharma Research Site, Yekaterinburg
- Spain (3):
  - Octapharma Research Site, Madrid
  - Octapharma Research Site, Oviedo
  - Octapharma Research Site, Santander
- Turkey (Türkiye) (5):
  - Octapharma Research Site, Antalya
  - Octapharma Research Site, Cebeci/Ankara
  - Octapharma Research Site, Fatih/Istanbul
  - Octapharma Research Site, Kazimdirik
  - Octapharma Research Site, Melikgazi/Kayseri

IPD SHARING:
Plan to Share IPD: No